CLINICAL TRIAL: NCT01583660
Title: Clinical Research of the Prognostic Influence of NSAIDS's Anti-inflammatory Effect on Senior Patients With Hip Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Army General Hospital (Other Government)
Responsible Party: Principal Investigator, Li Shaoguang, Li Shaoguang, Beijing Army General Hospital
Other Study IDs: EC-KS-2011-026
Record Dates: First submitted 2012-02-13; First posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Hip Fracture
Keywords: NSAIDs; Anti-inflammatory; elderly hip fracture; mortality
MeSH Terms: conditions — Hip Fractures | interventions — Celecoxib; oxycodone-acetaminophen; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood serum
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib — 200mg, PO.Bid, last from admission to hospital to one week after operation.
  Other Names: celebrex
Drug: Acetaminophen oxycodone — 1 tablet(Acetaminophen 325mg oxycodone 5mg), Q6h orally take,last from admission to hospital to one week after operation.
  Other Names: Oxydodone and Acetaminophen Tablets

SUMMARY:
With the development of society, aged population is growing. Hip fracture is the most common disease for aged people. With the life being longer than before, incidence of this disease is growing. The mortality of this disease is high-- almost 10% patients will die within 1 month, about 1/3 of patients will die within 12 months. About 20%-30% aged people who have hip fracture will die within one year.

The damaged organs caused by excessive inflammatory is one of possible reasons to cause higher mortality. Therefore, the investigators imagined that if they gave medicines to patients in time to reduce the inflammatory level, the inflammatory might have less effects on organs, and the recovery could be improved.

The investigators hypothesis on the basic research: the anti-inflammatory function of non steroidal antiinflammatory drugs (NSAIDs) can inhibit the inflammatory level of elderly hip fracture, so as to improve the recovery level and reduce the complicating disease and mortality. The investigators designed a clinic study to research NSAIDS' effects on inflammatory level and prognosis of elderly hip fracture.

DETAILED DESCRIPTION:
With the development of society, aged population is growing. The number of the aged people over 60 years old now reaches to 130 million. Hip fracture is the most common disease for aged people. According to Britain's statistical data of hip fracture, the average age of males who have hip fracture is 84 years old, and female, 83 years old, and female patients account for 74% of all the reported cases. The disease is deadly-- when attacked almost 10% patients die within 1 month, about 1/3 of patients die within 12 months. When seniors are attacked by hip fracture, about 20%-30% die within one year, 25% recover to normal life before the attack, and 55% patients become disabled in different degrees. Senile fracture has become an important issue relating to public health, brought huge burdens to average families. While developing very fast, our modern society has to come up with a solution to this urgent scientific problem.

The study has shown that the increasing inflammatory cytokines after senile fracture are independent dangerous factors of death and complications and the systemic inflammatory response after senile fracture causes organ damage and may explain why the seniors attacked by hip fracture are more likely to die than their peers. Therefore, we intend to give drug therapy to patients in the early stage after the attack, to reduce the inflammatory response of the body, thus reducing the damage of the body by the inflammatory response, and improving the prognosis of patients.

By inhibiting cyclooxygenase COX, and in turn the arachidonic acid (AA)'s transformation into prostaglandians (PGs) and thromboxane TXA, NSAIDs produces anti-inflammatory, antipyretic, analgesic and anti-rheumatism actions. It has been widely applied in clinic. According to study, there are two cyclooxygenase insomers in human body namely COX-1 and COX-2. COX-1, which exists in normal tissues, with physiological stimulation, can stimulate arachidonic acid to produce thromboxane A, prostaglandin e (PGE2) and prostacyclin I2 (PGI2). It can therefore protect the gastrointestinal tract, kidney, platelets, and vascular endothelial cells, and is also called structural enzyme. COX-2 is a type of COX induced by cytokines and produced under inflammatory stimulation, COX-2 mediates arachidonic acid to produce PGE-2 and PGI-2. As inflammatory prostaglandin, COX-2 has inflammation-causing effects and pain-causing effects. Its inhibition lays the pharmacological foundation for the antipyretic, analgesic, and anti-inflammatory effects of NSAIDs

Some animal experiment has showed that the inhibitor of COX-2 reduces the inflammatory expression of animal models after multiple severe traumas and enhances the survival rate. Recent reports suggest that the inhibitor of COX-2 (parecoxib) can reduce pro inflammatory cytokines after traumas, chemokine level and relieve acute lung injury. Clinic study shows that if applying the inhibitor of COX-2 into arthroplasty, the level of systemic inflammatory cytokines can be reduced, and a better postoperative function realized. There has been no report about the treatment of inflammatory response by NSAID after severe trauma.

In clinic, pain treatment has been conventional in modern wards and become a symbol of modern wards. In the newly published British NICE clinical guidelines of hip fracture, pain treatment of patients with hip fracture is pointed out as an appropriate method. Sufficient pain-treating enables patients to take part in necessary activities, and undergo medical examination, nursing care and rehabilitation. N-acethy aminophenol (paracetamol) is recommended. In case that the alone application of N-acethy aminophenol cannot completely relieve the pain, opiate drugs should be added. The guideline does not recommend NSAIDS since it may induce gastrointestinal complication. However, since it overcomes the side effect of gastrointestinal reaction, NSAIDS as a fundamental drug in pain treatment, especially an inhibitor of COX-2 has been widely applied in the treatment of trauma pain. But its anti-inflammatory effect has not been paid enough attention. Based on the above findings and research foundations, we wonder that besides its analgesic effect, whether NSAIDS has a equally beneficial anti-inflammatory effect on the excessive inflammatory response patient with severe trauma, and senior patients with hip fracture and improve their prognosis. Therefore, based on the fundamental research, we assume that the anti-inflammatory effect of NSAIDs can relieve the systemic inflammatory effect of senior patients with hip fracture, improve their prognosis, reduce incidence of complications and deaths. Through a prospective clinical experiment, we plan to study the effect of NSAIDS on the changes of inflammatory factors of senior patients with hip fracture, and their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* age > 60 years old,
* new patients with hip fracture(intertrochanteric fractures and femoral neck fractures),
* sign informed consent,
* can be followed up

Exclusion Criteria:

* have autoimmune disease,
* with blood disease, a history of thrombosis,
* with sulfonamides, aspirin or celebrex race Levin allergies,
* pathological fracture

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients(age > 60 years old)with hip fracture(intertrochanteric fractures and femoral neck fractures)adimited into Beijing Army General Hospital
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tiangsheng Sun, Prof., Study Chair — Beijing Army General Hospital
Locations (1):
- Beijing Army General Hospital, Beijing, Beijing Municipality, China